CLINICAL TRIAL: NCT02401620
Title: Validation of a Specific Questionnaire to Assess the Tolerability of the Different Therapeutic Strategies in Rheumatoid Arthritis
Brief Title: Validation of a Tolerability Questionnaire in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Antonio D Gómez-Centeno, MD, Corporacion Parc Tauli
Other Study IDs: FUN-TOC-2014-01
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: AR: arthritis rheumatoid; DMARDs: Disease-modifying antirheumatic drugs; ACR. American College of Rheumatology; EULAR: European League against rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single-group studies: Patients with RA diagnosed

SUMMARY:
The purpose of the present study is to assess the measurement properties of a tolerability questionnaire. The results obtained in patients with Rheumatoid Arthritis (RA) being treated will be robust and will assess the patient's tolerability to the treatment. Patients with greater tolerability will be more satisfied with their treatment.

DETAILED DESCRIPTION:
Clinicians do not have any standardized questionnaire to assess the tolerability from the patient's perspective. The tolerability assessment of the different pharmacological strategies for Rheumatoid Arthritis, from the patient's perspective, would provide additional information, improve doctor-patient communication and improve both adherence to and efficacy of treatment. For these reasons, the development and validation of a new tool is necessary not only for future researches, but for use in standard clinical practice.

The first phase of the development of the questionnaire has already been completed. The second phase of the development of the questionnaire has been designed at to validate the tool in the Spanish population.

This study aims to assess the measurement properties of a new tool which assesses the impact of daily life in Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old.
2. Patients with RA diagnosed according to the standards of the ACR (American College of Rheumatology) in 1987 or to the ACR/EULAR in 2010
3. Patients on treatment with any Rheumatoid Arthritis drug for at least 3 months before their inclusion in the study *
4. Patients who have provided informed consent prior to taking part in the study.

   * It's not necessary for patients to be treated in first-line at the moment of the inclusion in the study.

Exclusion Criteria:

1. Patients with rheumatic disease other than Rheumatoid Arthritis. Will be exclude patients with the following concomitant diseases: Rheumatic autoimmune disease other than RA; Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis; Diagnosis of juvenile idiopathic arthritis; inflammatory joint disease other than Rheumatoid Arthritis.
2. Patients with any other concomitant disease or treatment that, under clinical criteria, could affect the results of the study or any major episode of infection or disease requiring hospitalization.
3. Patients with any other medical or physiological condition that, in the view of the investigator, could compromise the ability of the patient to answer the study questions.
4. Patients who participated in interviews of the Phase I (development of the questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Rheumatoid Arthritis
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Validation of a new questionnaire to measure the tolerability to the pharmacological treatment in RA patients in patient's perspective. | 10 months
  To validate (evaluate measurement properties) a new questionnaire to measure the tolerability to the pharmacological treatment in RA patients in routine clinical practice

SECONDARY OUTCOMES:
the feasibility of the questionnaire by non-response rate and the time required to complete it | 10 months
  To assess the feasibility of the questionnaire by non-response rate and the time required to complete it
the construct validity of the questionnaire analyzing the relation between questionnaire scores and clinical data (discriminant validity). | 10 months
  To assess the construct validity of the questionnaire analyzing the relation between questionnaire scores and clinical data (discriminant validity
the reliability of the questionnaire in terms of internal consistency | 10 months
  To assess the reliability of the questionnaire in terms of internal consistency
describe socio-demographic and clinical features of the patients recruited in the study. | 10 months
  To describe socio-demographic and clinical features of the patients recruited in the study.
the adverse reactions (AR) reported by patients impact in the daily life. | 10 months
  To assess the adverse reactions (AR) reported by patients impact in the daily life
correlation between the tolerability questionnaire and the patient satisfaction | 10 months
  To assess the correlation between the tolerability questionnaire and the patient satisfaction (ARTS questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gomez Centeno, Study Chair — Hospital Corporacio Parc Tauli
Locations (6):
- Spain (6):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital Moisés Broggi, Sant Joan Despí, Barcelona
  - Hospital Can Misses, Ibiza Town, Ibiza
  - Hospital Son Espases, Mallorca, Mallorca
  - Hospital Son Llàtzer, Mallorca, Mallorca
  - Hospital Corporacio Sanitaria Parc Tauli, Sabadell, Spain